CLINICAL TRIAL: NCT04022824
Title: Vascular Responses After Percutaneous Coronary Intervention With Stenting In Patients With Obstructive Sleep ApNea: A Serial 3-Vessel Optical Coherence Tomography Study (VISION)
Brief Title: Vascular Responses After Percutaneous Coronary Intervention With Stenting In Patients With Obstructive Sleep Apnea
Acronym: VISION
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Shao-Ping Nie, Professor of Medicine, Director, Emergency & Critical Care Center, Beijing Anzhen Hospital
Other Study IDs: 2017034
Record Dates: First submitted 2019-07-01; First posted 2019-07-17 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Coronary Artery Disease; Obstructive Sleep Apnea of Adult
Keywords: Coronary artery disease; Obstructive sleep apnea; Optical coherence tomography; Vascular response
MeSH Terms: conditions — Coronary Artery Disease; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OSA
  Interventions: Other: OSA
- Non-OSA
  Interventions: Other: Non-OSA

INTERVENTIONS:
Other: OSA — Patients with OSA (apnea hypopnea index ≥15) based on sleep study
  Groups: OSA
Other: Non-OSA — Patients without OSA (apnea hypopnea index <15) based on sleep study
  Groups: Non-OSA

SUMMARY:
Obstructive sleep apnea (OSA) is an increasingly common chronic disorder in adults. Compared to the general population, OSA occurs more often in patients with coronary artery disease (CAD), with a reported prevalence of 38% to 65%. Emerging evidence indicates OSA initiates and exacerbates coronary atherosclerosis. Moreover, several observational studies indicate the presence of OSA was associated with higher rate of restenosis and repeat revascularization (mainly attributed non-culprit lesion revascularization) after percutaneous coronary intervention (PCI). OSA might initiate endothelial injury by repetitive bursts of sympathetic activity that occur with apneas and hypopneas. Moreover, untreated OSA reduces endothelial repair capacity. Whether OSA could exacerbate neointimal proliferation and plaque progression in the non-culprit lesion after drug-eluting stent (DES) implantation remains less studied. The investigators aimed to evaluate neointimal proliferation and strut coverage within stent segment as well as changes of plaque volume and morphology in the non-culprit lesion by optical coherence tomography (OCT) in patients with versus without OSA at 12-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 80 years old
2. Patients undergoing PCI with stenting in at least one de novo lesion in a native coronary artery
3. 3-vessel OCT was available visually (at least one pullback/vessel)
4. Written informed consent

Exclusion Criteria:

1. Predominantly central sleep apnea (CSA, ≥50% central events or central apnea hypopnea index ≥10/h)
2. Previous or current use of continuous positive airway pressure (CPAP)
3. Cardiogenic shock (systolic arterial pressure <90mmHg), congestive heart failure (NYHA or Killip≥3)
4. STEMI within 1 week
5. Prior PCI or CABG
6. Chronic kidney disease [eGFR<60ml/(min*1.73m2)]
7. Aortic-coronary ostial lesion
8. Left main lesion
9. Chronic total occlusion
10. In-stent restenotic lesion
11. A tortuous vessel and/or severely calcified lesion or severe stenosis and the OCT catheter could not pass across the lesion
12. Massive residual thrombus on angiography despite thrombus aspiration or thrombectomy
13. Planned elective PCI within 12 months
14. Severe comorbidities: eg. malignancy (life expectancy <2 years)
15. Known or planned pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing PCI with stenting and 3-vessel OCT and receiving overnight sleep study (polygraphy)
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2018-04-18 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Relative proliferation volume within stent segment (% of stent volume) | 12 months

SECONDARY OUTCOMES:
Change of total lipid volume index in the non-culprit lesion | 12 months
Maximum area stenosis within stent segment | 12 months
  Defined as minimal lumen area divided by the mean of reference lumen area
Total proliferation volume within stent segment | 12 months
Maximum proliferation area within stent segment | 12 months
Minimal lumen area within stent segment | 12 months
Prevalence of uncovered struts, uncovered and apposed struts, malapposed struts | 12 months
Prevalence of neoatherosclerosis | 12 months
Total lipid volume index | Baseline
  Defined as the averaged lipid angle multiplied by lipid length; including culprit and non-culprit lesions
Prevalence of TCFA | Baseline
  In the culprit and non-culprit lesions
Prevalence of plaque rupture | Baseline
  In the culprit and non-culprit lesions
Rate of major adverse cardiac events (cardiac death, myocardial infarction, or ischemic-driven repeat revascularization) | 12 months

OTHER OUTCOMES:
Maximum lipid angle | Baseline
Calcium volume | Baseline
Macrophage volume | Baseline
Correlation of total lipid volume index with AHI | Baseline
Correlation of total lipid volume index with lowest SpO2 | Baseline
Correlation of total lipid volume index total time with SpO2 <90% | Baseline
Total lipid volume index stratified by sex in both groups | Baseline
Total lipid volume index stratified by obesity in both groups | Baseline
Total lipid volume index stratified by diabetes in both groups | Baseline
Rate of individual cardiovascular events | 12 months
  Including all-cause death, cardiac death, myocardial infarction, target vessel revascularization, target lesion revascularization, non-target vessel revascularization, hospitalization for unstable angina

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Capital Medical University, Beijing, China